CLINICAL TRIAL: NCT01160783
Title: Genetic Contributions to Autism Spectrum Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Walsh, Chief, Division of Genetics & Genomics, Boston Children's Hospital
Other Study IDs: 07-04-0136
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Autism; Asperger's Syndrome; Pervasive Developmental Disorder
Keywords: Autism; Asperger's Syndrome; Asperger Syndrome; Autistic Disorder; Autism Spectrum Disorder; Pervasive Developmental Disorders; Pervasive Developmental Disorder-Not Otherwise Specified; Child Development Disorders, Pervasive; PDD-NOS
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, DNA and RNA and/or Saliva, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is working towards gaining a better understanding of the genetic and environmental factors involved in autism spectrum disorders (ASD), which includes autism, pervasive developmental disorder (PDD), and Asperger's syndrome. The investigators hope that information gained from this study will lead to new ways of diagnosing and treating ASDs.

DETAILED DESCRIPTION:
Participation generally takes less than 2 hours to complete and travel to Children's Hospital Boston is not required. Participants are asked some questions about their medical and family history. The investigators also request permission to review medical records related to the ASD diagnosis. Finally, the investigators obtain a small blood or saliva sample in order to search for genes that may be important in understanding ASD. The investigators can arrange for the blood draw through a participant's physician or a clinical laboratory and saliva samples can be obtained through the mail. The study questions are answered via telephone or mailed questionnaires. There is no cost to participate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an Autism Spectrum Disorder (autism, pervasive developmental disorder (PDD), or Asperger's syndrome)
* Age > 18 months

Exclusion Criteria:

* Do not have the diagnosis of an ASD
* Participation in the "Phenotypic and Genetic Risk Factors in ASD" study at Boston Children's Hospital.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with a diagnosis of an Autism Spectrum Disorder (autism, pervasive developmental disorder (PDD), or Asperger's syndrome) and their parents and/or siblings
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2007-04; Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Gene expression levels | At sample collection
  Gene expression levels

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Walsh, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No